CLINICAL TRIAL: NCT00310414
Title: fMRI Studies of Task Specificity in Focal Hand Dystonia
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060128; 06-N-0128
Record Dates: First submitted 2006-03-31; First posted 2006-04-03 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2012-03-13

CONDITIONS: Focal Dystonia
Keywords: Imaging Studies; Botulinum Toxin; Writer's Cramp; Focal Hand Dystonia; FHD; Writer Cramp; Healthy Volunteer; HV
MeSH Terms: conditions — Dystonic Disorders; Dystonia, Focal, Task-Specific

SUMMARY:
This study will examine how the brain makes involuntary spasms and contractions in patients with focal hand dystonia (FHD). Patients with dystonia have muscle spasms that cause uncontrolled twisting and repetitive movement or abnormal postures. In FHD, only the hand is involved. The study will use functional magnetic resonance imaging (fMRI, see below) to study which areas of the brain are primarily affected in FHD and better understand how brain changes produce dystonia symptoms.

Normal right-handed volunteers and patients with FHD who are 18-65 years of age may be eligible for this study. Candidates are screened with a medical history and physical and neurological examinations. Women who can become pregnant have a urine pregnancy test.

All participants undergo fMRI. This test uses a strong magnetic field and radio waves to obtain images of body organs and tissues. The subject lies on a table that is moved into the scanner (a metal cylinder), wearing earplugs to muffle loud knocking and thumping sounds that occur during the scanning process. The procedure lasts about 90 minutes, during which time the patient is asked to lie still for 10-15 minutes at a time. During the procedure, subjects are asked to perform some tasks, including writing, tapping with their hand, and drawing in a zigzag motion. Each task is performed using the right hand, left hand and right foot.

DETAILED DESCRIPTION:
Objective:

Writer's cramp, a form of focal hand dystonia, is the most frequently observed task specific dystonia. Symptoms of writer's cramp often appear as soon as the pen is picked up, or after a few words of writing. Patients with simple writer's cramp have difficulties writing, but carry out other tasks with the affected hand without spasms. Little is known about why the hand spasms when writing, while performing other tasks normally.

The purpose of this study is to identify brain areas of activation associated specifically with the task of handwriting with the dystonic hand, in patients with simple writer's cramp. Simple writer's cramp can be defined by a patient exhibiting the symptoms only when writing and symptoms are not present in any other task performance. Specifically for this study, patients should be able to write for 20 seconds consecutively in a run. We plan to use functional magnetic resonance imaging (fMRI) to identify the pattern of blood oxygenation level-dependent (BOLD) activation in the brain when different tasks are performed by different limbs in healthy volunteers and patients with focal hand dystonia.

Study Population:

This research will be conducted using 22 patients diagnosed with simple writer's cramp and 32 healthy volunteers matched for age and gender.

Design:

Using a block design in functional magnetic resonance imaging (fMRI), we will examine the brain activity of patients and healthy volunteers while they execute three tasks: writing, tapping and a zigzagging motion, with three separate limbs: the dystonic hand, the opposite hand, and the right foot.

Outcome Measures:

The changes in signal intensity of the brain activity correlated with the motor program (task of handwriting) and effector (dystonic hand) will be collected and analyzed.

The findings we expect to obtain with this experiment may contribute to basic knowledge of the linkage between task specificity and the dystonic hand, and may provide a better understanding of the pathophysiology of writer's cramp.

ELIGIBILITY:
* INCLUSION CRITERIA:

Focal Dystonia Subjects must be:

* Right hand dominant
* Between 18 and 65 years old
* Diagnosed with mild, simple focal hand dystonia. For this study mild, simple focal hand dystonia suggests that the patient does not present symptoms when performing tasks other than writing. Additionally, the patient should be able to write for 20 seconds consecutively
* Willing to abstain from alcohol 48 hours prior to the study

Volunteers must be:

* Healthy right-handed dominant individuals
* Between 18 and 65 years old
* Willing to abstain from alcohol 48 hours prior to the study

EXCLUSION CRITERIA:

* Subjects with implanted devices such as pacemakers, medication pumps or defibrillators, metal in the cranium except mouth, intracardiac lines, history of shrapnel injury or any other condition/device that may be contraindicated or prevent the acquisition of MRI
* Subjects with any finding on the MRI safety questionnaire which prevents them from safely undergoing an MRI scan
* Subjects who are pregnant.
* Subjects with claustrophobia or other restrictions which prevent them from undergoing a scan in a confined space for up to 60 minutes
* Subjects with any visual, motor, or hearing difficulties
* Subjects with severe focal hand dystonia i.e., subjects who experience dystonic spasms in tasks other than/in addition to writing
* Subjects with mirror dystonia
* Subjects without the capacity to give consent
* Subjects with any history of a severe medical condition, such as cardiovascular disease, which will prevent them from lying flat for up to 60 minutes.
* Subjects with any history of brain tumor, stroke, head trauma or vascular malformation as obtained by history or from imaging studies.
* Subjects who have had recent (within 3 months) Botulinum Toxin (Botox) injections.
* Subjects who are on anti-parkinsonian drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2006-03-30; Study Completion 2012-03-13

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth H Fischbeck, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Berardelli A, Rothwell JC, Hallett M, Thompson PD, Manfredi M, Marsden CD. The pathophysiology of primary dystonia. Brain. 1998 Jul;121 ( Pt 7):1195-212. doi: 10.1093/brain/121.7.1195. PMID 9679773
- [Background] Butterworth S, Francis S, Kelly E, McGlone F, Bowtell R, Sawle GV. Abnormal cortical sensory activation in dystonia: an fMRI study. Mov Disord. 2003 Jun;18(6):673-82. doi: 10.1002/mds.10416. PMID 12784271
- [Background] Blood AJ, Flaherty AW, Choi JK, Hochberg FH, Greve DN, Bonmassar G, Rosen BR, Jenkins BG. Basal ganglia activity remains elevated after movement in focal hand dystonia. Ann Neurol. 2004 May;55(5):744-8. doi: 10.1002/ana.20108. PMID 15122718